CLINICAL TRIAL: NCT05627570
Title: Investigating the Effects of Diets With Different Types of Food Processing Following UK dietAry Guidance on healTh outcomEs: an 8-week Community-based Crossover Randomised Controlled Trial in People With Overweight or Obesity, Followed by a 6-month Behavioural Intervention
Brief Title: A Study Comparing the Health Effects of Two Diets Following UK Dietary Guidance in People Living With Overweight or Obesity
Acronym: UPDATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 151582
Record Dates: First submitted 2022-11-11; First posted 2022-11-25 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Cardiometabolic Syndrome; Overweight
Keywords: Food processing; Diet; Healthy, balanced diet; Dietary guidelines; Obesity; Cardiometabolic disease
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Overweight

STUDY DESIGN:
Intervention Model Description: 2x2, randomised, controlled crossover trial
Who Masked: Participant
Masking Description: To minimise unnecessary unblinding, participants will not be informed of the order in which they receive their diets, but it will likely become clear which diet they are consuming, and thus the study will not be considered to be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diet A then Diet B, followed by a 6-month behavioural support programme (Experimental): 8-weeks of Diet A then 8-weeks of Diet B, then 6 months of goal-based behavioural support for consuming a healthy, balanced diet, increasing physical activity and reducing sedentary behaviour.
  Interventions: Dietary Supplement: Healthy, balanced Diet A; Dietary Supplement: Healthy, balanced Diet B; Behavioral: Behavioural support intervention
- Diet B then Diet A, followed by a 6-month behavioural support programme (Experimental): 8-weeks of Diet B then 8-weeks of Diet A, then 6 months of goal-based behavioural support for consuming a healthy, balanced diet, increasing physical activity and reducing sedentary behaviour.
  Interventions: Dietary Supplement: Healthy, balanced Diet A; Dietary Supplement: Healthy, balanced Diet B; Behavioral: Behavioural support intervention

INTERVENTIONS:
Dietary Supplement: Healthy, balanced Diet A — Healthy, balanced diet following Eatwell Guide recommendations
Dietary Supplement: Healthy, balanced Diet B — Healthy, balanced diet following Eatwell Guide recommendations
Behavioral: Behavioural support intervention — Participants will work with a behavioural scientist to create a personal plan to eat a healthier diet and be more physically active. This support will last for 6 months, with ongoing monthly telephone/video calls with the research team.

SUMMARY:
There are two parts to this study:

1. The investigators will study if the benefit from eating a healthy, balanced diet depends on the types of food processing in the diet. The investigators will do this by providing participants with two diets that follow the Eatwell Guide (referred to in this study as Diet A and Diet B to avoid unblinding), but containing foods with different types of food processing, for 8 weeks each. The investigators will collect data on blood pressure, body composition, physical activity and fitness, questions regarding quality of life, mental health and wellbeing, and blood samples at the start of each diet and at 4 and 8 weeks into each diet.
2. The investigators will then study whether participants are able to switch from their usual unhealthy diet to a healthy, balanced diet, and the benefits of doing so. The investigators will do this by providing participants with 6 months of personal support. The investigators will also look at what helps participants to maintain a healthy diet, and what makes it difficult. The investigators will also support participants to be more physically active.

DETAILED DESCRIPTION:
Eating a healthy, balanced diet is important for health. A healthy, balanced diet involves eating a variety of foods in the right proportions. In the UK, the Eatwell Guide gives recommendations on what people should eat more of, and what people should eat less of. Unhealthy diets contain lots of foods high in saturated fat, added sugar and salt, which increases the risk of developing obesity, cardiovascular disease and type 2 diabetes. Advice for a healthy, balanced diet includes consuming five portions of fruit and vegetables per day and eating more high fibre foods. Following the healthy, balanced diet advice given in the Eatwell Guide can reduce the risk of poor health.

However, there are other parts of the diet that are not covered in the Eatwell Guide that may also be important for health. For example, research suggests that different types of food processing might influence health, but these types of food processing are not included within the recommendations.

It is unknown if the benefits of following the healthy diet advice in the Eatwell Guide depend on the types of food processing in the diet. It is important to find out if these types of food processing matter, in order to give people the best advice possible. It also means that the government and other health organisations may need to change the regulations around the food that people eat.

To answer this, the investigators will compare the effects of two healthy, balanced diets following the advice in the UK Eatwell Guide, but each based on a different type of food processing (referred to in this study as Diet A and Diet B to avoid unblinding). Participants will receive the first diet for 8 weeks, return to their normal diet for 4 weeks, and then receive the second diet for a further 8 weeks. Participants will have 6 months of support to help improve their diet and be more physically active. Participants will work with a behavioural scientist to create a personal plan to eat a healthier diet and be more physically active, using behaviour change techniques based on capability, opportunity, motivation - behaviour (COM-B) theory of behaviour change. This support will last for 6 months, with ongoing monthly telephone/video calls with the research team. The results from this study will be used to help inform UK dietary guidance and food policy.

There are two parts to this study:

1. The investigators will study if the benefit from eating a healthy, balanced diet depends on the types of food processing in the diet. The investigators will do this by providing participants with two diets (Diet A and Diet B) that follow the Eatwell Guide, but containing foods with different types of processing, for 8 weeks each.
2. The investigators will then study whether participants are able to switch from their usual unhealthy diet to a healthy, balanced diet, and the benefits of doing so. The investigators will do this by providing participants with 6 months of personal support. The investigators will also look at what helps participants to maintain a healthy diet, and what makes it difficult. The investigators will also support participants to be more physically active.

ELIGIBILITY:
Inclusion Criteria:

* Staff at University College London Hospitals (UCLH)
* Adults aged between [18 and 65] years old.
* BMI ≥25 kg/m2 (living with overweight or obesity)
* Weight stable for the past 3 months (≤5 % variation in body weight over preceding 3 months)
* Have a habitual dietary intake high in unhealthy food
* Able to read and write in English.
* Medically safe to participate in a dietary intervention programme.
* Willing and able to give written informed consent.
* Able to attend the relevant in person and online sessions.
* Able to comply with the study protocol (including dietary recommendations for each intervention and reporting adherence).
* Females of childbearing potential and males agree to use an effective method of contraception from the time consent is signed until the end of the intervention period and final follow-up assessment. Effective methods of contraception acceptable for this trial are outlined in Appendix 2.
* Females of childbearing potential must be on highly effective contraception and have a negative pregnancy test within 7 days of being randomised. NOTE: Participants are considered not of childbearing potential if they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.

Exclusion Criteria:

* Contraindication for dietary intervention
* Participation in another clinical intervention trial
* Concomitant usage of medications that cause weight gain or weight loss
* Cardiometabolic comorbidities (e.g. diabetes, on insulin)
* Coeliac disease
* Inflammatory bowel disease
* A diagnosed eating disorder
* Planning a weight management programme in the next 3 months
* Any diagnosed food allergy, or other allergies which limit the ability to adhere to the intervention diet
* Dietary restrictions (e.g. vegan or vegetarian) which limit the ability to adhere to the interventions
* BMI >40 kg/m2 or basal metabolic rate ≥2300/kcal/day (to ensure intervention diets are at least 300kcal/day greater than maintenance energy needs).
* Females who are pregnant, breast-feeding, or intends to become pregnant.
* A history of drug or alcohol abuse
* Any other factor making the participant unsuitable in the view of investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Mean difference in percent weight change (%WC) at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  %WC will be calculated using: %WC = ((weight at baseline - weight at timepoint after baseline)/weight at baseline) x 100, calculated at each intervention endpoint. Mean difference in percent weight change will be calculated as: percent weight change diet A - percent weight change diet B. Weight measured in kilograms.

SECONDARY OUTCOMES:
Changes in waist circumference at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using a tape measure
Changes in waist circumference after 6-months of the behavioural support programme | First baseline to 6-months follow-up
  Assessed using a tape measure
Changes in fat-free mass at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using bioelectrical impedance analysis (BIA)
Changes in fat-free mass after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using bioelectrical impedance analysis (BIA)
Changes in fat mass at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using bioelectrical impedance analysis (BIA)
Changes in fat mass after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using bioelectrical impedance analysis (BIA)
Changes in heart rate at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using an oximeter
Changes in heart rate after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using an oximeter
Changes in systolic and diastolic blood pressure at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using a sphygmomanometer
Changes in systolic and diastolic blood pressure after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using a sphygmomanometer
Changes in comorbidities at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Comorbidities assessed using medical records, physical examination and blood sample analyses
Changes in Liver function at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Fasted Liver function assessed using blood sample analyses
Changes in Glucose at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Fasted Glucose assessed using blood sample analyses
Changes in Lipids at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Fasted Lipids assessed using blood sample analyses
Changes in HbA1c at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Fasted HbA1c assessed using blood sample analyses
Changes in C-reactive protein (CRP) at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Fasted CRP assessed using blood sample analyses
Changes in metabolomics at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Fasted and fed metabolomics assessed using blood sample analyses
Changes in Comorbidities after 6-months of the behavioural support | First baseline to 6-months follow-up
  Comorbidities assessed using medical records, physical examination and blood sample analyses
Changes in Liver function after 6-months of the behavioural support | First baseline to 6-months follow-up
  Fasted Liver function assessed using blood sample analyses
Changes in Glucose after 6-months of the behavioural support | First baseline to 6-months follow-up
  Fasted Glucose assessed using blood sample analyses
Changes in metabolomics after 6-months of the behavioural support | First baseline to 6-months follow-up
  Fasted and fed metabolomics assessed using blood sample analyses
Changes in Lipids after 6-months of the behavioural support | First baseline to 6-months follow-up
  Fasted Lipids assessed using blood sample analyses
Changes in HbA1c after 6-months of the behavioural support | First baseline to 6-months follow-up
  Fasted HbA1c assessed using blood sample analyses
Changes in C-reactive protein (CRP) after 6-months of the behavioural support | First baseline to 6-months follow-up
  Fasted CRP assessed using blood sample analyses
Changes in appetite at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Fasted and fed appetite scores (Visual analogue scale) assessed using a meal test
Changes in gut hormones at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Fasted and fed circulating gut hormones assessed using a meal test
Changes in adipocytokines at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Fasted adipocytokines assessed using a meal test
Changes in appetite after 6-months of the behavioural support | First baseline to 6-months follow-up
  (a) Fasted and fed appetite scores (Visual analogue scale, 10 point scale, higher score indicates greater hunger) assessed using a meal test
Changes in gut hormones after 6-months of the behavioural support | First baseline to 6-months follow-up
  Fasted and fed circulating gut hormones assessed using a meal test
Changes in adipocytokines after 6-months of the behavioural support | First baseline to 6-months follow-up
  Fasted adipocytokines assessed using a meal test
Changes in sleep at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Change in objectively reported sleep assessed using accelerometry.
Changes in sleep quality at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Change in subjectively reported sleep assessed using the Pittsburgh Sleep Quality Index
  The Pittsburgh Sleep Quality Index is a validated 19-item measure, which will be used to determine sleep quality in the past month, to distinguish between good and poor sleepers. A higher score indicates poorer sleep quality.
Changes in sleep after 6-months of the behavioural support | First baseline to 6-months follow-up
  Change in objectively reported sleep assessed using accelerometry.
Changes in sleep quality after 6-months of the behavioural support | First baseline to 6-months follow-up
  Change in subjectively reported sleep assessed using the Pittsburgh Sleep Quality Index
  The Pittsburgh Sleep Quality Index is a validated 19-item measure, which will be used to determine sleep quality in the past month, to distinguish between good and poor sleepers. A higher score indicates poorer sleep quality.
Changes in physical activity at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  (a) Change in objectively reported physical activity levels (sedentary, light (LPA), moderate (MPA), vigorous (VPA)) assessed using accelerometry
Changes in physical activity levels at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Change in subjectively reported physical activity levels (sedentary, light (LPA), moderate (MPA), vigorous (VPA)) assessed using the short form International Physical Activity Questionnaire (IPAQ-SF).
  The short-form International Physical Activity Questionnaire (IPAQ-SF) is a standardised questionnaire consisting of 7 questions that ask about physical activity in the past 7 days. IPAQ-SF will be used to subjectively assess time spent in light, moderate and vigorous physical activity levels, and time spent sitting. The questionnaire takes a few minutes to complete. Higher physical activity values indicate greater physical activity levels, higher time spent sitting indicates greater sedentary behaviour.
Changes in physical activity after 6-months of the behavioural support | First baseline to 6-months follow-up
  (a) Change in objectively reported physical activity levels (sedentary, light (LPA), moderate (MPA), vigorous (VPA)) assessed using accelerometry
Changes in physical activity levels after 6-months of the behavioural support | First baseline to 6-months follow-up
  Change in subjectively reported physical activity levels (sedentary, light (LPA), moderate (MPA), vigorous (VPA)) assessed using the short form International Physical Activity Questionnaire (IPAQ-SF).
  The short-form International Physical Activity Questionnaire (IPAQ-SF) is a standardised questionnaire consisting of 7 questions that ask about physical activity in the past 7 days. IPAQ-SF will be used to subjectively assess time spent in light, moderate and vigorous physical activity levels, and time spent sitting. The questionnaire takes a few minutes to complete. Higher physical activity values indicate greater physical activity levels, higher time spent sitting indicates greater sedentary behaviour.
Changes in handgrip strength at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using a hand dynamometer.
Changes in handgrip strength after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using a hand dynamometer.
Changes in walking distance at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using the 6-minute walk test (6MWT)
Changes in changes in walking distance after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using the 6-minute walk test (6MWT)
Changes in leg strength at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using the sit-to-stand (STS) test
Changes in leg strength after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using the sit-to-stand (STS) test
Changes in quality of life at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using EuroQoL 5 dimensions 3 levels (EQ-5D-3L)
  EQ-5D-3L is a 6-item self-reported questionnaire that consists of a descriptive system to assess the following 5 domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression using 3 levels (e.g. mobility: I have no problems walking about, I have some problems walking about, or I am confined to bed, higher score indicates worse quality of life) and a visual analogue scale, which records self-rated health on a 0 to 100 scale (100 = best health).
Changes in quality of life after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using EuroQoL 5 dimensions 3 levels (EQ-5D-3L)
  EQ-5D-3L is a 6-item self-reported questionnaire that consists of a descriptive system to assess the following 5 domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression using 3 levels (e.g. mobility: I have no problems walking about, I have some problems walking about, or I am confined to bed, higher score indicates worse quality of life) and a visual analogue scale, which records self-rated health on a 0 to 100 scale (100 = best health).
Changes in weight-related quality of life at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using Impact of Weight on Quality of Life-Lite (IWQOL-Lite)
  Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a 31-item, self-reported, obesity and overweight-specific measure of health-related quality of life. This tool consists of a total score, scoring on five aspects - physical function, self-esteem, sexual life, public distress, and work. Higher scores indicate a better quality of life.
Changes in weight-related quality of life after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using Impact of Weight on Quality of Life-Lite (IWQOL-Lite)
  Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a 31-item, self-reported, obesity and overweight-specific measure of health-related quality of life. This tool consists of a total score, scoring on five aspects - physical function, self-esteem, sexual life, public distress, and work. Higher scores indicate a better quality of life.
Changes in mental wellbeing at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS)
  The Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) is a 14-item, positively worded, validated measure of mental wellbeing, with 5 responses, which are summed to produce a single measure of wellbeing. Scores range from 14 to 70, with higher scores indicating greater positive mental wellbeing.
Changes in mental wellbeing after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS)
  The Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) is a 14-item, positively worded, validated measure of mental wellbeing, with 5 responses, which are summed to produce a single measure of wellbeing. Scores range from 14 to 70, with higher scores indicating greater positive mental wellbeing.
Changes in depression at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using Patient Health Questionnaire-9 (PHQ-9)
  The Patient Health Questionnaire (PHQ-9) is a 9-item validated measure, which will be used to assess the severity of depression. Each item is rated from 0 to 3, for a total score out of 27. A score of 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Changes in depression after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using Patient Health Questionnaire-9 (PHQ-9)
  The Patient Health Questionnaire (PHQ-9) is a 9-item validated measure, which will be used to assess the severity of depression. Each item is rated from 0 to 3, for a total score out of 27. A score of 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Changes in anxiety at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using Generalised Anxiety Disorder Assessment-7 (GAD-7)
  The Generalised Anxiety Disorder assessment (GAD-7) is a 7-item anxiety scale, which will be used to screen and measure the severity of generalised anxiety disorder. Each item is rated from 0 to 3, for a total score out of 21. A score of 11-15 indicates moderately severe anxiety, and 16-21 of severe anxiety.
Changes in anxiety after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using Generalised Anxiety Disorder Assessment-7 (GAD-7)
  The Generalised Anxiety Disorder assessment (GAD-7) is a 7-item anxiety scale, which will be used to screen and measure the severity of generalised anxiety disorder. Each item is rated from 0 to 3, for a total score out of 21. A score of 11-15 indicates moderately severe anxiety, and 16-21 of severe anxiety.
Changes in eating behaviour (psychological impact of living in food-abundant environments) at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using Power of Food scale
  The Power of Food (PoF) scale is a 15-item validated measure, which will be used to assess the psychological impact of living in food-abundant environments. Higher scores indicate greater psychological impact of living in a food-abundant environment
Changes in eating behaviour (psychological impact of living in food-abundant environments), after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using Power of Food scale
  The Power of Food (PoF) scale is a 15-item validated measure, which will be used to assess the psychological impact of living in food-abundant environments. Higher scores indicate greater psychological impact of living in a food-abundant environment
Changes in eating behaviour (severity and type of food cravings) at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using Control of Eating Questionnaire
  The Control of Eating Questionnaire (CoEQ) is a 21-item validated measure, which will be used to measure the severity and type of food cravings. Higher scores indicate greater agreement with the statement (severity and type of food cravings)
Changes in eating behaviour (severity and type of food cravings), after 6-months of the behavioural support | First baseline to 6-months follow-up
  Assessed using Control of Eating Questionnaire
  The Control of Eating Questionnaire (CoEQ) is a 21-item validated measure, which will be used to measure the severity and type of food cravings. Higher scores indicate greater agreement with the statement (severity and type of food cravings)
(In a subset of participants) Changes in brain functional resting state connectivity at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Assessed using functional brain magnetic resonance imaging and diffusion weighted imaging.
(In a subset of participants) Changes in brain functional resting state metabolism at 8 weeks between Diet A and Diet B | Baseline to 8 weeks for both diets
  Metabolite changes assessed using magnetic resonance spectroscopy.
Changes in aspects of behaviour regulation after 6-months of the behavioural support programme | First baseline to 6-months follow-up (49 weeks)
  (a) Barriers and facilitators to healthy eating and physical activity, assessed using a capability, opportunity, motivation - behaviour (COM-B) questionnaire
  Participants will complete one questionnaire investigating the barriers and facilitators to physical activity and healthy eating, based on the COM-B model of behaviour change. The survey contains 257 items; the physical activity component contains 137 items, and the eating component contains 120 items.This survey is expected to take 30 minutes. The survey uses a range of items (Likert scale, yes/no, agree/disagree, true/false) with levels of agreement yes/no indicating barriers or facilitators to behaviour.
Barriers and facilitators to eating a healthy, balanced diet | 6-months follow-up
  Assessed using a one to one semi-structured telephone/video call interview at 6-months follow-up
  The aim of the qualitative interviews is to gain an in-depth understanding of the barriers and facilitators to adherence to a minimally processed diet, and to map these onto an intervention development framework. Interviews will follow a simple topic guide designed to explore motivations for participating and experiences of the trial, with a particular focus on barriers and facilitators to adhering to a minimally processed diet.
  The qualitative process will use Framework Analysis and other methods of thematic analysis designed to explore experiences of a behaviour change trials.
Changes in diet after 6-months of the behavioural support programme | First baseline to 6-months follow-up
  (a) Changes in food and nutrient intake, assessed using 24-hour recall (Intake24)
  24-hour recalls will be conducted using Intake24, a validated, online, self-reported dietary recall system, based on a multiple-pass 24-hour recall that is suitable for the general population (https://intake24.co.uk). The recall takes on average 12 minutes to complete58. The system is self-completed and will guide the participant through the recall process. Firstly, the user will list all food and drink consumed, followed by probing questions about quantity consumed and further information on food and drink reported.
Changes in habitual diet after 6-months of the behavioural support programme | First baseline to 6-months follow-up
  (a) Changes in food and nutrient intake, assessed using food frequency questionnaire (FFQ) (European Prospective Investigation of Cancer (EPIC)-Norfolk FFQ)
  Food frequency questionnaires can be used to determine average food intakes over longer durations of time. Average food intakes will be assessed using the European Prospective Investigation into Cancer and Nutrition (EPIC)-Norfolk FFQ, a validated, semi-quantitative measure of average dietary intake over the past year.
  The EPIC-Norfolk FFQ is split into two sections, part 1 contains a 130-item food list. Each item contains an individual food, combination of individual foods or a food type. Participants tick the most appropriate frequency of consumption of that food item from nine options (from never or less than once per month, to 6+ per day). Part 2 asks more detailed questions relating to the food items in part 1, including types of fats used in cooking, types of milks consumed and choice of cereals.
Changes in weekly food shopping expenditure at 6-months follow-up will be compared with the first baseline, based on changes in reported dietary intakes | First baseline to 6-months follow-up
  Assessed using 24-hour recall (Intake24)
  24-hour recalls will be conducted using Intake24, a validated, online, self-reported dietary recall system, based on a multiple-pass 24-hour recall that is suitable for the general population (https://intake24.co.uk). The recall takes on average 12 minutes to complete58. The system is self-completed and will guide the participant through the recall process. Firstly, the user will list all food and drink consumed, followed by probing questions about quantity consumed and further information on food and drink reported.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Batterham, Professor, Principal Investigator — UCL, UCL Hospitals
Locations (1):
- UCL, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heuchan GN, Buck C, Conway R, Dicken S, Brown AC, Jassil FC, Makaronidis J, Van Tulleken C, Gandini Wheeler-Kingshott CA, Batterham R, Fisher A. Development, content and planned evaluation of a behavioural support intervention to reduce ultraprocessed food intake and increase physical activity in UK healthcare workers: UPDATE trial stage 2 study protocol. BMJ Open. 2025 Oct 29;15(10):e107435. doi: 10.1136/bmjopen-2025-107435. PMID 41161844
- [Derived] Dicken SJ, Jassil FC, Brown A, Kalis M, Stanley C, Ranson C, Ruwona T, Qamar S, Buck C, Mallik R, Hamid N, Bird JM, Brown A, Norton B, Gandini Wheeler-Kingshott CAM, Hamer M, van Tulleken C, Hall KD, Fisher A, Makaronidis J, Batterham RL. Ultraprocessed or minimally processed diets following healthy dietary guidelines on weight and cardiometabolic health: a randomized, crossover trial. Nat Med. 2025 Oct;31(10):3297-3308. doi: 10.1038/s41591-025-03842-0. Epub 2025 Aug 4. PMID 40760353
- [Derived] Dicken S, Makaronidis J, van Tulleken C, Jassil FC, Hall K, Brown AC, Gandini Wheeler-Kingshott CAM, Fisher A, Batterham R. UPDATE trial: investigating the effects of ultra-processed versus minimally processed diets following UK dietary guidance on health outcomes: a protocol for an 8-week community-based cross-over randomised controlled trial in people with overweight or obesity, followed by a 6-month behavioural intervention. BMJ Open. 2024 Mar 11;14(3):e079027. doi: 10.1136/bmjopen-2023-079027. PMID 38471681